CLINICAL TRIAL: NCT06340048
Title: Epicardial Injection of Allogeneic Human Pluripotent Stem Cell-derived Cardiomyocytes to Treat Severe Chronic Ischemic Heart Failure
Brief Title: Epicardial Injection of hiPSC-CMs to Treat Severe Chronic Ischemic Heart Failure
Acronym: HEAL-AHF
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Help Therapeutics (Industry)
Collaborators: TEDA International Cardiovascular Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: XC Liu
Record Dates: First submitted 2024-01-15; First posted 2024-04-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2025-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HiCM-188 Low dose therapy (Experimental): Intramyocardial injection of HiCM-188 (50 million) during CABG surgery.
  Interventions: Drug: HiCM-188 therapy
- HiCM-188 Medium dose therapy (Experimental): Intramyocardial injection of HiCM-188 (150 million) during CABG surgery.
  Interventions: Drug: HiCM-188 therapy
- HiCM-188 High dose therapy (Experimental): Intramyocardial injection of HiCM-188 (450 million) during CABG surgery.
  Interventions: Drug: HiCM-188 therapy

INTERVENTIONS:
Drug: HiCM-188 therapy — Epicardial Injection of Allogeneic Human Pluripotent Stem Cell-derived Cardiomyocytes (HiCM-188) during coronary artery bypass grafting surgery

SUMMARY:
The purpose of this clinical study is to evaluate the feasibility, safety and efficacy of intramyocardial injection of human induce pluripotent stem cell-derived cardiomyocytes (HiCM-188) during coronary artery bypass grafting (CABG) surgery in patients with severe chronic ischemic heart failure.

DETAILED DESCRIPTION:
This is a single center, open-label, three-group dose-escalation (phase I) study followed by dose-extension (phase IIa) study in up to 36 severe ischemic heart failure patients. It is estimated that up to 18 phase I patients will be received HiCM-188 intramyocardial injection during CABG surgery. The maximum number of subjects after dose escalation and dose extension studies in each dose group is 12. All the subjects need take immunosuppressant after transplantation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Willingness and ability to give written informed consent
3. Nuclide-myocardial metabolic perfusion imaging or Magnetic Resonance Imaging (MRI) revealed infarcted myocardium in the left anterior descending branch (LAD) coronary artery supply area
4. LVEF<50% as assessed by Echocardiography or LVEF≤40% as assessed by MRI
5. Patients have indications for Coronary Artery Bypass Grafting

Exclusion Criteria:

1. Presence of a pacemaker, implantable cardioverter-defibrillator (ICD), or cardiac resynchronization therapy device (CRT)
2. Diagnosed with malignancy within 5 years
3. Autoimmune disease
4. Recipients of organ transplant.
5. Patients undergoing other surgical operations (excluding resection of ventricular aneurysm and left atrial appendage excision/occlusion).
6. Severe ventricular arrhythmia
7. Contraindication to CABG surgery
8. Contraindication to cardiac MRI or PET/CT scan.
9. Contraindication to immunosuppressants
10. Participation in another clinical trial within 3 months prior to screening
11. Pregnancy, lactation, or a positive serum pregnancy test
12. Any other condition considered by the investigator to be inappropriate for inclusion in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2026-11-10 (Estimated); Study Completion 2027-05-10 (Estimated)

PRIMARY OUTCOMES:
The incidence of major Serious Adverse Events (SAE) | Within the first month after surgery
  The incidence of major Serious Adverse Events (SAE) within the first month after surgery, including pericardial tamponade, nonfatal myocardial infarction, stroke, and all-cause death

SECONDARY OUTCOMES:
Grade 4 or above arrhythmias Related to HiCM-188 Cell Therapy | Within the first month after surgery
  Grade 4 or above arrhythmias associated with the HiCM-188 therapy within the first month after surgery
The incidence of tumor | 12 months after surgery
  assessed by PET whole-body imaging at baseline and 12 months after HiCM-188 therapy
Left ventricular geometry as assessed by cardiac magnetic resonance imaging (MRI) | Baseline, 6 and 12 months after surgery
  Left ventricular wall thickness, interventricular septum thickness
Size of myocardial infarction as assessed by MRI | Baseline, 6 and 12 months after surgery
  Size of myocardial infarction
Ventricular wall motion as assessed by MRI | Baseline, 6 and 12 months after surgery
  Ventricular wall motion
Left ventricular ejection fraction as assessed by MRI | Baseline, 6 and 12 months after surgery
  Left ventricular ejection fraction
Cardiac Volumes as assessed by MRI | Baseline, 6 and 12 months after surgery
  Left ventricular end-diastolic volume (LVEDV), Left ventricular end-systolic volume (LVESV) and Stroke Volume (SV)
Cardiac output (CO) as assessed by MRI | Baseline, 6 and 12 months after surgery
  Cardiac output (CO)
End-diastolic myocardial mass as assessed by MRI | Baseline, 6 and 12 months after surgery
  End-diastolic myocardial mass
Left ventricular ejection fraction (LVEF) as assessed by Echocardiography | Baseline, 6 and 12 months after surgery
  Left ventricular ejection fraction
Fractional shortening (FS) as assessed by Echocardiography | Baseline, 6 and 12 months after surgery
  Fractional shortening
Left ventricular dimensions as assessed by Echocardiography | Baseline, 6 and 12 months after surgery
  Left ventricular end-diastolic diameter (LVEDD), left ventricular end-systolic diameter(LVESD)and left atrial diameter
Cardiac Volumes as assessed by Echocardiography | Baseline, 6 and 12 months after surgery
  Left ventricular end- diastolic volume (LVEDV) and Left ventricular end-systolic volume(LVESV)
Mitral valve inflow spectrum(E/A) as assessed by Echocardiography | Baseline, 6 and 12 months after surgery
  Mitral valve inflow spectrum (E/A)
Longitudinal strain as assessed by Echocardiography | Baseline, 6 and 12 months after surgery
  Longitudinal strain
Myocardial viability as assessed by SPECT | Baseline, 6 and 12 months after surgery
  Myocardial viability
Myocardial blood flow as assessed by SPECT | Baseline, 6 and 12 months after surgery
  Myocardial blood flow
NT-proBNP Levels | Baseline, 6 and 12 months after surgery
  The changes of NT-proBNP Levels
6-minute walking distance | Baseline, 6 and 12 months after surgery
  The changes of 6-minute walking distance at 6M and 12M after HiCM-188 therapy
New York Heart Association (NYHA) functional classification | Baseline, 6 and 12 months after surgery
  The changes of New York Heart Association (NYHA) functional classification at 6M and 12M after HiCM-188 therapy
Changes of Quality of Life (QoL) as assessed by Minnesota Living with Heart Failure Questionnaire (MLHFQ) | Baseline, 6 and 12 months after surgery
  The MLHFQ is a self-administered disease-specific outcome measure instrument for patients with heart failure (HF), comprising 21 items rated on Likert scales, representing different degrees of impact of HF on QoL.
  The MLHFQ scores are on a range of 0-105, in which higher scores reflect better health status.
Changes of Quality of Life(QOL) as assessed by 36-Item Short Form Survey (SF-36) | Baseline, 6 and 12 months after surgery
  The 36-Item Short Form Survey(SF-36) is a self-administered outcome measure instrument that comprises 36 items grouped into 8 dimensions: limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems, limitations in usual role activities because of physical health problems, bodily pain, general mental health, limitations in usual role activities because of emotional problems, vitality, general health perceptions.
  The SF-36 scores are on a range of 0-100, in which higher scores reflect better health status.

CONTACTS AND LOCATIONS:
Locations (1):
- TEDA International Cardiovascular Hospital, Tianjin, Tianjin Municipality, China